CLINICAL TRIAL: NCT03743610
Title: Investigation of Physiological Adaptations to Simulated Intermittent Altitude on Human Health and Performance
Brief Title: Physiological Adaptations to Simulated Intermittent Altitude on Human Health and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney M. Wheatley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-000484
Record Dates: First submitted 2018-11-12; First posted 2018-11-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Altitude Hypoxia
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Effect of heart rate training in simulated altitude (Experimental): Participants will exercise in simulated altitude start at a minimum of 2,000ft and will increase to no greater than 16,400ft with each visit. The increase will be in accordance to maintaining >65% max heart rate during room air based maximal peak work.
  Interventions: Other: Simulated altitude
- Effect of saturation of oxygen training in simulated altitude (Experimental): Participants will exercise in simulated altitude start at a minimum of 2,000ft and will increase to no greater than 16,400ft with each visit. The increase will be in accordance to maintaining 40-60% of max work rate during room air work rate and based upon saturation of oxygen of between 70-80%.
  Interventions: Other: Simulated altitude
- Effect of optimized training in simulated altitude (Active Comparator): Participants will perform the more beneficial intervention (heart rate or saturation of oxygen training) to evaluate whether it improves elite athlete's training status at altitude.
  Interventions: Other: Simulated altitude
- Effect of placebo training in non-simulated altitude (Placebo Comparator): Participants will perform placebo beneficial intervention (heart rate or saturation of oxygen training) to evaluate whether the optimized protocol truely improves elite athlete's training status at altitude.
  Interventions: Other: Placebo simulated altitude

INTERVENTIONS:
Other: Simulated altitude — Participants will exercise in simulated altitude will range between 2100 feet and 16400 feet and will increase according to arm guidelines
  Arms: Effect of heart rate training in simulated altitude; Effect of optimized training in simulated altitude; Effect of saturation of oxygen training in simulated altitude
Other: Placebo simulated altitude — Participants will exercise at sea level at similar percentage of intensities to the simulated altitude group.
  Arms: Effect of placebo training in non-simulated altitude

SUMMARY:
The investigators expect to find that different intensity and altitude exposure levels will show what kind of intermittent exposure protocol is more beneficial to athletes and healthy individuals that experience acute exposure to altitude during exercise. This may furthermore be related to acute altitude exposure for recreational exercise use as well.

ELIGIBILITY:
Inclusion criteria:

* 18-70 years of age,
* history of good health,
* generally active to competitive athletes.

Exclusion criteria:

* History of cardiac or pulmonary disease,
* not currently active,
* unable to exercise or meet study requirements (e.g., number of sessions),
* live at altitude (>2,100m or 7,000ft).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | Baseline, 2-week, 4-week, 6-week, and 8-week
Change in hematocrit | Baseline, 2-week, 4-week, 6-week, and 8-week
Change in erythropoietin | Baseline, 2-week, 4-week, 6-week, and 8-week

SECONDARY OUTCOMES:
Change in peak VO2 | Baseline and 6- and 8-week
  Change from maximal exercise test performed at sea level
Change in cycling performance at altitude | Baseline and 6- and 8-week
  change in aerobic/anaerobic cycling performance at altitude

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Wheatley, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials